CLINICAL TRIAL: NCT02191553
Title: Differential Effect of Four Mindfulness Exercises on Mindfulness, Cerebral Cartography and Heart Ratio Variability
Brief Title: Differential Effect of Four Mindfulness Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, PhD, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI13/0129
Record Dates: First submitted 2014-07-09; First posted 2014-07-16 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Well-being; Depression; Anxiety
Keywords: mindfulness meditation; alpha rhythm; EEG; brain mapping; emotion; attention
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Whole Body Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Group: Relaxation Techniques (Active Comparator): Relaxation techniques which do not involve either formal or informal mindfulness training. Subjects in this group practice Jacobson's progressive muscular relaxation, emotional imagining and Schultz's autogenic training.
  Interventions: Behavioral: Control group relaxation techniques
- Loving Kindness Meditation (Metta) (Experimental): Loving-kindness meditation following Kristin Neff protocol
  Interventions: Behavioral: Loving-kindness meditation
- Body Scan (Experimental): Body scan as described in standard MBSR protocol
  Interventions: Behavioral: Body scan
- Sitting Practice (Experimental): Sitting practice as mindfulness meditation described in standard MBSR protocols.
  Interventions: Behavioral: Sitting practice

INTERVENTIONS:
Behavioral: Control group relaxation techniques — Jacobson's progressive muscular relaxation, emotional imagining and Schultz's autogenic training.
  Arms: Control Group: Relaxation Techniques
Behavioral: Loving-kindness meditation — Following Kristin Neff protocol
  Arms: Loving Kindness Meditation (Metta)
Behavioral: Body scan — Body scan: Attention being directed with detailed awareness to every part of the body for a sustained period of time.
  Arms: Body Scan
Behavioral: Sitting practice — In the sitting exercise, participants are guided to pay attention to a certain range of still points, starting with attention to breathing. In this exercise attention is fully concentrated on a single object: the sensation attached to breathing. If the mind wanders or is distracted by an external stimulus, attention is gently returned to sensations derived from breathing.
  Arms: Sitting Practice

SUMMARY:
Mindfulness can be considered as a family of complex attentional and emotional regulation strategies that promote the cultivation of well-being and emotional balance. The practice of mindfulness produces the development of a consciousness that unfolds moment to moment, open and unprejudiced in the present moment, here and now. Despite its extensive benefits, the practice of mindfulness requires a significant commitment in time and effort, which limits the potential for its dissemination. The studies to narrow the differential effects of the various exercises based on mindfulness, will further enhance their effectiveness and they can guide the practice sequence according to user needs. In this paper we will research mindfulness electroencephalographic correlates of as four different exercise programs included in mindfulness-based cognitive therapy (MBCT) and stress reduction program based on mindfulness (MBSR) as well as its effect on several psychological variables.

DETAILED DESCRIPTION:
Mindfulness is a way of using attention intentionally, repeatedly reactivating the attentional focus, so that it enhances the ability of sustained attention. It involves a complex process of self-regulation and inhibition of internal and external stimuli interferences.

Although the overall effects of meditation on brain bioelectrical signals are still being characterized, there is some consensus on the fact that meditation helps alter brain activity in both state and trait.

The specific aim of this study is to assess the differential effect of four different practices of mindfulness in psychological well-being and their corresponding neurophysiological correlates.

The hypothesis is that different exercises within the range of mindfulness practices exert different effects in terms of electroencephalographic activity, expecting different band increases in alpha (activity 7-to 2 Hz), beta (activity more than 13 Hz), theta (activity 4-6 Hz) and delta (activity less than 3 Hz) respectively, as well as changes in the lateralization of the activity (left or right hemisphere). We also expect an improvement in the variables such as mindfulness, self-compassion, positive affect, anxiety, depression and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* sign of informed consent
* no previous meditation training experience

Exclusion Criteria:

* mental or neurologic disorder
* respiratory disease
* previous brain damage history
* medication intake that could interfere in the electroencephalographic results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Different facets of Mindfulness | 3 months
  The Five Facets Mindfulness Questionnaire (FFMQ) will be used: It assesses the following facets of mindfulness: Observing, describing, acting with awareness, non judging of inner experience and non-reactivity to inner experience

SECONDARY OUTCOMES:
Brain function | 3 months
  We will use cerebral cartography
Positive and negative affectivity | 3 months
  It will be measured with PANAS questionnaire
anxiety and depression | 3 months
  Measured with Hospital Anxiety Depression Scale
Insomnia | 3 months
  Measured with Pittsburgh Sleep Quality Index (PSQI)
Self-compassion | 3 months
  Measured with Self-Compassion Scale

OTHER OUTCOMES:
heart function and heart variability rate | 3 months
  The investigators will use electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Javier García Campayo, Dr, Principal Investigator — Aragon Health Sciences Institute (IACS)
Locations (1):
- Arrabal Health Center, Zaragoza, Spain

REFERENCES:
- [Background] Soler J, Cebolla A, Feliu-Soler A, Demarzo MM, Pascual JC, Banos R, Garcia-Campayo J. Relationship between meditative practice and self-reported mindfulness: the MINDSENS composite index. PLoS One. 2014 Jan 22;9(1):e86622. doi: 10.1371/journal.pone.0086622. eCollection 2014. PMID 24466175
- [Background] Fayed N, Lopez Del Hoyo Y, Andres E, Serrano-Blanco A, Bellon J, Aguilar K, Cebolla A, Garcia-Campayo J. Brain changes in long-term zen meditators using proton magnetic resonance spectroscopy and diffusion tensor imaging: a controlled study. PLoS One. 2013;8(3):e58476. doi: 10.1371/journal.pone.0058476. Epub 2013 Mar 25. PMID 23536796